CLINICAL TRIAL: NCT06980402
Title: Pragmatic Pilot Study of SKH@Home Post-discharge Monitoring Initiative on Outcomes of Surgical Patients
Brief Title: Post-discharge Monitoring Initiative on Outcomes of Post-surgical Patients
Acronym: SKH@home
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sengkang General Hospital (Other)
Responsible Party: Principal Investigator, Chue Koy Min, Consultant, Clinical Assistant Professor, Department of General Surgery, Sengkang General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-4580
Record Dates: First submitted 2025-02-20; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Laparoscopy; Discharge Planning
Keywords: Bariatric surgery; Laparoscopic surgery; Abdominal abscesses; Liver abscesses; Discharge planning
MeSH Terms: conditions — Abdominal Abscess; Liver Abscess | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard inpatient care until deemed suitable for discharge (Active Comparator): Post-surgical patients are routinely monitored in the acute hospital setting, until they are deemed suitable for discharge by their primary surgeon.
  Interventions: Procedure: Standard inpatient care until deemed suitable for discharge
- Early post-surgical discharge with post-surgical home based monitoring (Experimental): The SKH@home program, is a post-discharge monitoring program, which allows stable post-surgical patients (after minimally invasive/ endoscopic/ bariatric surgery) or with stable surgical conditions after interventions (like abdominal or liver abscess management) to be discharged earlier from the acute hospital while providing regular post-discharge monitoring at the patient's own home, either through home visits or patient assessment via telemonitoring.
  Interventions: Procedure: Early post-surgical discharge with post-surgical home based monitoring

INTERVENTIONS:
Procedure: Early post-surgical discharge with post-surgical home based monitoring — The SKH@home program, is a post-discharge monitoring program, which allows stable post-surgical patients to be discharged earlier from hospital while providing regular post-discharge monitoring at the patient's own home, either through home visits and patient assessment, or telemonitoring of patients.
  Arms: Early post-surgical discharge with post-surgical home based monitoring
Procedure: Standard inpatient care until deemed suitable for discharge — Patients will receive standard postoperative management in the acute hospital until they are deemed fit for discharge by their primary surgeon
  Arms: Standard inpatient care until deemed suitable for discharge

SUMMARY:
The investigators are conducting a prospective study to evaluate the SKH@Home programme, a post-discharge monitoring initiative for surgical patients. The aim of this study is to conduct a pragmatic, non-randomized pilot study to compare the SKH@Home programme with standard post-surgical care on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is keen for home management
2. Hemodynamically stable
3. Able and willing to self-care and monitor / Good social support
4. Lives in Singapore's Northeast region

   EITHER
5. Diagnosed with intra-abdominal abscess requiring ongoing IV antibiotics as recommended by Infectious Diseases Specialist where necessary OR Diagnosed with liver abscess requiring ongoing IV antibiotics as recommended by Infectious Diseases Specialist where necessary AND Has undergone initial treatment (e.g., drainage if required) and is clinically improving

   OR
6. Underwent an uneventful straightforward bariatric surgical procedure, and has been monitored overnight without any immediate postoperative issues OR Underwent uneventful straightforward laparoscopic/ endoscopic/ minimally invasive surgery, and has been monitored for at least 6 hours without any immediate postoperative issues AND has no significant intraprocedural concerns by the operating surgeon

Exclusion Criteria:

1. Unable to self-care / no caregiver
2. Requires daily review by the surgical team
3. Suspicion of surgical complications requiring surgical intervention
4. Requires post-discharge monitoring care for > 2 weeks
5. Unregulated psychiatric disorders
6. Daily flushing of drains required

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Bed days saved | From enrollment to 30 days after patient is discharged from the hospital/ post-discharge monitoring programme
  Bed days saved in the acute hospital setting
Return to hospital | From enrollment until 30-days after patient is discharged from the hospital/ from post-discharge monitoring care
  Unplanned readmission/ return to the hospital within 30-days
Length of stay | From enrollment until patient is discharged from the hospital/ from post-discharge monitoring care (up to around 2 weeks), whichever is longer
  Combined length of stay. For inpatients, will be time of admission till time of discharge from acute hospital For patients enrolled into post-discharge monitoring programme, will be from time of admission till time of discharge from post-discharge monitoring programme
Hospitalisation bill | From enrollment until 30-days after patient is discharged from the hospital/ from post-discharge monitoring care
  Total non-subsidised hospitalisation bill size
Postoperative complications | From enrollment until 30-days after patient is discharged from the hospital/ from post-discharge monitoring care
  30-day postoperative complications, graded by the Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Koy Min Chue, Principal Investigator — Sengkang General Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McGillion MH, Parlow J, Borges FK, Marcucci M, Jacka M, Adili A, Lalu MM, Ouellette C, Bird M, Ofori S, Roshanov PS, Patel A, Yang H, O'Leary S, Tandon V, Hamilton GM, Mrkobrada M, Conen D, Harvey V, Lounsbury J, Mian R, Bangdiwala SI, Arellano R, Scott T, Guyatt GH, Gao P, Graham M, Nenshi R, Forster AJ, Nagappa M, Levesque K, Marosi K, Chaudhry S, Haider S, Deuchar L, LeBlanc B, McCartney CJL, Schemitsch EH, Vincent J, Pettit SM, DuMerton D, Paulin AD, Simunovic M, Williams DC, Halman S, Harlock J, Meyer RM, Taylor DA, Shanthanna H, Schlachta CM, Parry N, Pichora DR, Yousuf H, Peter E, Lamy A, Petch J, Moloo H, Sehmbi H, Waggott M, Shelley J, Belley-Cote EP, Devereaux PJ; PVC-RAM-1 Investigators. Post-discharge after surgery Virtual Care with Remote Automated Monitoring-1 (PVC-RAM-1) technology versus standard care: randomised controlled trial. BMJ. 2021 Sep 30;374:n2209. doi: 10.1136/bmj.n2209. PMID 34593374
- [Result] Gunter RL, Chouinard S, Fernandes-Taylor S, Wiseman JT, Clarkson S, Bennett K, Greenberg CC, Kent KC. Current Use of Telemedicine for Post-Discharge Surgical Care: A Systematic Review. J Am Coll Surg. 2016 May;222(5):915-27. doi: 10.1016/j.jamcollsurg.2016.01.062. Epub 2016 Feb 13. No abstract available. PMID 27016900
- [Result] Jonker LT, Lahr MMH, Oonk MHM, de Bock GH, van Leeuwen BL. Post-discharge Telemonitoring of Physical Activity, Vital Signs, and Patient-Reported Symptoms in Older Patients Undergoing Cancer Surgery. Ann Surg Oncol. 2021 Oct;28(11):6512-6522. doi: 10.1245/s10434-021-09707-3. Epub 2021 Feb 27. PMID 33641013
- [Result] van Ede ES, Scheerhoorn J, Buise MP, Bouwman RA, Nienhuijs SW. Telemonitoring for perioperative care of outpatient bariatric surgery: Preference-based randomized clinical trial. PLoS One. 2023 Feb 22;18(2):e0281992. doi: 10.1371/journal.pone.0281992. eCollection 2023. PMID 36812167
- [Result] Cooper S, Patel S, Wynn M, Provost D, Hassan M. Outcomes of same-day discharge in bariatric surgery. Surg Endosc. 2024 Sep;38(9):5122-5129. doi: 10.1007/s00464-024-11053-w. Epub 2024 Jul 19. PMID 39028346